CLINICAL TRIAL: NCT07401784
Title: Efficacy and Safety Evaluation of Remote Ischemic Adaptation ( Intermittent Pressure Stimulation ) in the Treatment of Insomnia After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-I-2025-045
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Apoplexy; Depression Anxiety Disorder; Cerebrovascular Disease
Keywords: Remote ischemic adaptation technology; cerebral apoplexy; Depression Anxiety Disorder; Cerebrovascular Disease
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- treatment group (Experimental): The full-automatic ischemic preconditioning therapeutic instrument was used to pressurize the patients ' upper arms ( experimental group pressure = 200 mmHg ) for 5 minutes, and then breathe out for 5 minutes, which was an ischemia-reperfusion cycle. Each training was performed for 5 consecutive cycles, once in the morning and once in the afternoon, twice a day, at least 5 days a week, for a total of 4 weeks.
  Interventions: Device: Automatic ischemic preconditioning therapeutic apparatus
- control group (Sham Comparator): Participants in this group will use a sham training device that is identical in appearance, sound, and sense of wear to the experimental device. The treatment plan was consistent with the experimental group in time and process : wearing a cuff for 5 minutes, rest for 5 minutes, a total of 5 cycles. The key difference is that during the so-called ' pressure ', the cuff is inflated to a pressure of only 60 mmHg to simulate the sense of operation of the device and a slight sense of skin contact. The treatment frequency, cycle and execution personnel were the same as those of the experimental group.
  Interventions: Device: Sham Ischemic Preconditioning Device

INTERVENTIONS:
Device: Automatic ischemic preconditioning therapeutic apparatus — The patient 's upper arms were pressurized for 5 minutes( Test group pressure = 200 mmHg ), and then breathed for 5 minutes. It was an ischemia-reperfusion cycle. Each training was performed for 5 consecutive cycles, 1 in the morning and 1 in the afternoon, 2 times / day, at least 5 days a week, for a total of 4 weeks.
  Arms: treatment group
Device: Sham Ischemic Preconditioning Device — A sham training device that is identical in appearance, sound, and wear sensation to the experimental device. During the "pressure" phase, the cuff is inflated to a non-ischemic low pressure (60 mmHg) to mimic device operation. The treatment schedule (cycles, frequency, duration) is identical to the experimental arm.
  Arms: control group

SUMMARY:
The incidence of post-stroke depression is high, which will affect the rehabilitation of neurological function, damage cognitive function, and increase the risk of subsequent stroke recurrence. The guidelines recommend that in addition to antiplatelet, blood pressure control, lipid-lowering and other treatments, secondary prevention of post-stroke depression should also be strengthened. Moreover, after the occurrence of post-stroke depression, methods such as medication and psychotherapy have their own limitations, such as potential adverse drug reactions and limited psychotherapy. Therefore, it is necessary to pay attention to the prevention of post-stroke depression.

The remote ischemic adaptation therapy applied in our study is a safe, non-invasive and convenient physical therapy. By transiently and repeatedly applying ischemia-reperfusion stimulation to both upper arms, it induces a systemic protective response, improves the brain 's tolerance to ischemia and hypoxia, and exerts a protective effect on multiple organs such as the brain and heart. The RIC therapeutic instrument has been national patented and has been maturely applied to the prevention and treatment of acute cerebral infarction, which can promote the rehabilitation of neurological function. In addition, it also has certain curative effect in the treatment of cerebrovascular stenosis, refractory hypertension, depression, insomnia, anxiety and so on.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and one of the main causes of disability. The incidence of stroke is increasing worldwide. In 2010, the number of patients with first stroke increased by 68 % compared with 1990. The long-term effects of stroke sequelae include mobility, cognitive ability, language and communication disorders, as well as emotional problems, difficulties in daily life activities and social barriers. Sleep often changes after stroke. Insomnia disorder is a risk factor for stroke and an independent predictor of life satisfaction 6 months after stroke. Insomnia disorder is a sleep disorder characterized by frequent and persistent difficulty in falling asleep and / or difficulty in maintaining sleep and leading to poor sleep quality. Insomnia disorder can exist in isolation or co-exist with mental disorders, physical diseases or substance abuse, which can be accompanied by a variety of functional impairments during awakening. It is reported that in the general population, the prevalence of insomnia is 6 % to 48 % according to different definitions of insomnia. The prevalence of insomnia is higher in stroke patients. Insomnia after stroke has a high correlation with depression, disability and fatigue, and has a greater impact on returning to work one year after stroke. Therefore, actively dealing with the insomnia symptoms of stroke patients is conducive to improving the prognosis of stroke patients and improving the quality of life of stroke patients. The current treatment methods are divided into drug therapy and non-drug therapy. Drug therapy mainly includes benzodiazepines and barbiturates, but its clinical application and long-term use are limited due to many adverse reactions, contraindications, and strong dependence. In addition to drug therapy, other treatments for post-stroke depression and insomnia include psychotherapy, strong light therapy, transcranial magnetic stimulation and acupuncture. Some evidence shows that these methods are beneficial to the improvement of insomnia, fatigue, mood and quality of life, but the conclusions are different and the quality of evidence is low.

Remote ischemic condition ( RIC ), also known as intermittent pressure stimulation, is a non-invasive and easy-to-use physical therapy that has been used in clinical trials to protect the brain ( including ischemic and hemorrhagic stroke ), heart and many other organs. Studies have shown that RIC also has the effect of treating depression, insomnia and anxiety, but the research reports on the treatment of insomnia after stroke are still limited. At present, the mechanism of insomnia after stroke is unknown, and there may be many factors involved, such as inflammatory stress, stroke location, environmental factors, etc. The potential mechanisms of RIC include anti-inflammatory, anti-oxidative stress, immune system regulation and other potential pathways. Therefore, RIC can be used as a promising non-invasive physical therapy for post-stroke insomnia.

Therefore, this study takes patients with post-stroke insomnia as the research object, uses RIC technology to treat patients with post-stroke insomnia, and observes its therapeutic effect and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old ;
* In line with the diagnostic criteria of ischemic stroke, with reference to the ' Chinese guidelines for the diagnosis and treatment of acute ischemic stroke ' diagnosed ischemic stroke ;
* Despite adequate sleep opportunities, patients still have difficulty in falling asleep or maintaining sleep, staying asleep at least 3 times a week for at least 3 months, which leads to pain or impaired daytime function.
* PSQI score ≥ 6 and ISI score ≥ 8 ;
* All research contents have been understood and informed consent has been signed.

Exclusion Criteria:

* Insomnia before stroke ;
* Patients with mental disorders, bipolar disorder or depression, generalized anxiety disorder and other mental disorders ;
* Patients were pregnant or lactating women ;
* Other reasons identified by the researchers are not suitable for patients ;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency as measured by polysomnography | 4 weeks
  Sleep efficiency is calculated as (total sleep time / total time in bed) × 100%, assessed by overnight polysomnography. Higher percentage indicates better sleep efficiency.
Insomnia Severity Index (ISI) total score | 4 weeks
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing perceived insomnia severity. Each item is rated on a 0-4 scale, yielding a total score ranging from 0 to 28. Higher scores indicate more severe insomnia.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) global score | 4 weeks, 3 months, 6 months
  he PSQI is a self-rated questionnaire assessing sleep quality over the past month. It contains 19 items generating 7 component scores, which are summed to yield a global score ranging from 0 to 21. Higher scores indicate worse sleep quality.
Change from baseline in sleep onset latency (SOL) as measured by polysomnography | 4 weeks
  Sleep onset latency is defined as the time from lights out to the first epoch of any stage of sustained sleep (in minutes), measured by overnight polysomnography. The change from baseline to post-intervention will be calculated. Lower values indicate faster sleep onset.
Change from baseline in total sleep time (TST) as measured by polysomnography | 4 weeks
  Total sleep time is the total duration of all sleep stages (N1, N2, N3, REM) during the recording night (in minutes), measured by overnight polysomnography. The change from baseline to post-intervention will be calculated. Higher values indicate longer sleep duration.
Change from baseline in percentage of stage N1 sleep (N1%) as measured by polysomnography | 4 weeks
  Stage N1 sleep is the transitional, lightest stage of non-rapid eye movement (NREM) sleep. N1% is calculated as (total time in N1 sleep / total sleep time) × 100%, derived from overnight polysomnography. The change from baseline to post-intervention will be calculated.
Change from baseline in percentage of stage N2 sleep (N2%) as measured by polysomnography | 4 weeks
  Stage N2 sleep is a stable stage of NREM sleep characterized by sleep spindles and K-complexes. N2% is calculated as (total time in N2 sleep / total sleep time) × 100%, derived from overnight polysomnography. The change from baseline to post-intervention will be calculated.
Change from baseline in percentage of stage N3 sleep (N3%) as measured by polysomnography | 4 weeks
  Stage N3 sleep is deep sleep or slow-wave sleep. N3% is calculated as (total time in N3 sleep / total sleep time) × 100%, derived from overnight polysomnography. The change from baseline to post-intervention will be calculated. Higher values typically indicate more deep sleep.
National Institutes of Health Stroke Scale (NIHSS) total score | 4 weeks, 3 months, 6 months
  The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. It assesses level of consciousness, gaze, visual fields, facial palsy, motor strength, ataxia, sensation, language, dysarthria, and extinction/inattention. The total score ranges from 0 (no deficit) to 42 (severe deficit). A lower score indicates less severe neurological impairment.
modified Rankin Scale (mRS) score | 4 weeks, 3 months, 6 months
  The mRS is a clinician-reported measure of global disability in patients with stroke. It is a single-item scale ranging from 0 to 6: 0 (No symptoms), 1 (No significant disability), 2 (Slight disability), 3 (Moderate disability), 4 (Moderately severe disability), 5 (Severe disability), 6 (Death). A lower score indicates better functional outcome.
Barthel Index (BI) score | 4 weeks,3 months,6 months
  The Barthel Index is an ordinal scale used to measure performance in basic activities of daily living (ADL), including feeding, bathing, grooming, dressing, bowel and bladder control, toileting, chair transfer, ambulation, and stair climbing. The total score ranges from 0 (fully dependent) to 100 (fully independent) . A higher score indicates greater independence in ADL.
Functional Independence Measure (FIM) total score | 4 weeks,3months,6months
  The Functional Independence Measure is a standardized assessment of functional independence used in rehabilitation settings. It measures the level of assistance a person requires to perform basic life activities. The scale comprises 18 items covering two domains: Motor (13 items) and Cognitive (5 items). Each item is scored from 1 (total assistance) to 7 (complete independence). The total score ranges from 18 (totally dependent) to 126 (completely independent). A higher score indicates a greater level of functional independence.
Mini-Mental State Examination (MMSE) total score | 4 weeks,3months,6months
  The MMSE is a brief 30-point questionnaire used to screen for cognitive impairment. It assesses orientation, registration, attention and calculation, recall, language, and visual construction. The total score ranges from 0 to 30, with a higher score indicating better cognitive function. A score below 24 is typically indicative of cognitive impairment.
Montreal Cognitive Assessment (MoCA) total score | 4 weeks,3 months,6 months
  The MoCA is a cognitive screening tool designed to detect mild cognitive impairment. It assesses multiple domains: visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. The total score ranges from 0 to 30, with a higher score indicating better cognitive function. A score of 26 or above is generally considered normal.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT07401784/Prot_SAP_000.pdf